CLINICAL TRIAL: NCT00089921
Title: A 24-Week, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study of the Efficacy of Oral SCIO-469 in Subjects With Active Rheumatoid Arthritis Who Are Not Receiving DMARDs Other Than Hydroxychloroquine
Brief Title: SPRiNG: SCIO-469 Patients With Rheumatoid Arthritis Not Receiving Methotrexate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Scios, Inc. (Industry)
Responsible Party: VP CLINICAL RESEARCH, Centocor Research & Development, Inc., PA, USA
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005167; SCIO-469ARA2003; B007
Record Dates: First submitted 2004-08-17; First posted 2004-08-20 (Estimated); Last update posted 2010-10-18 (Estimated); Status verified 2010-10

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid Arthritis; DMARDs; Methotrexate; p38 kinase
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — SCIO-469

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 001 (Experimental): SCIO-469 30 mg capsule three times daily for 12 weeks
  Interventions: Drug: SCIO-469
- 002 (Experimental): SCIO-469 60 mg capsule three times daily for 12 weeks
  Interventions: Drug: SCIO-469
- 003 (Experimental): SCIO-469 100 mg tablet once daily for 12 weeks
  Interventions: Drug: SCIO-469
- 004 (Placebo Comparator): Placebo 2 capsules three times daily and one tablet daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SCIO-469 — 60 mg capsule three times daily for 12 weeks
  Arms: 002
Drug: SCIO-469 — 30 mg capsule three times daily for 12 weeks
  Arms: 001
Drug: Placebo — 2 capsules three times daily and one tablet daily
  Arms: 004
Drug: SCIO-469 — 100 mg tablet once daily for 12 weeks
  Arms: 003

SUMMARY:
The primary objective of this study is to determine the efficacy of oral SCIO-469 in patients with rheumatoid arthritis who are not receiving liver damaging (hepatotoxic) disease-modifying anti-rheumatic drugs (DMARDs).

DETAILED DESCRIPTION:
This is a 24 week randomized (study drug assigned by chance), double blind (neither physician nor patient knows the name of the assigned drug), placebo controlled, parallel group study assessing the safety and effectiveness of oral SCIO-469 in treating patients with rheumatoid arthritis who are not receiving liver damaging (hepatotoxic) disease-modifying anti-rheumatic drugs (DMARDs). The patient will participate in the study for approximately 183 days. Safety measures will include vital signs (blood pressure, pulse rate, breathing rate), 12-lead electro-cardiogram, adverse events, concomitant medications, and clinical laboratory evaluations (including serum chemistry, hematology, qualitative urinalysis, and liver function tests). The patient may be assigned to receive 30 mg capsule orally (by mouth) as one or two capsules three times daily, or receive 100 mg tablet orally once daily, or placebo (no active drug) orally as two capsules three times daily and placebo tablet orally once daily for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients having active rheumatoid arthritis who are not receiving medications known as hepatotoxic disease-modifying anti-rheumatic drugs (DMARDs)
* Patients taking hydroxychloroquine (Plaquenil) must be on a stable or consistent dose prior to entering study

Exclusion Criteria:

* Patients using Enbrel, Remicade, Kineret, Humira, or an experimental biologic agent within the past 3 months
* Lab tests revealed elevated liver enzymes within the past 6 months
* Medical history of Tuberculosis, cancer, multiple sclerosis, neuropathy or encephalopathy
* HIV positive
* Abnormal electrocardiogram
* Chronic or acute infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2004-07; Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
ACR20 is 20% reduction in tender and swollen joint counts and 20% improvement in three of the five remaining ACR core set measures: patient and physician global assessments, visual analog scale for pain, HAQ, and an acute-phase reactant (CRP or ESR) | Day 1 to approximately Day 85 of treatment

SECONDARY OUTCOMES:
ACR50 responders at Week 12 | 12 weeks
ACR20 and ACR50 responders at each evaluation visit other than Week 12 | 24 weeks
All individual variables of the ACR response criteria at each evaluation visit | 24 weeks
Disease Activity Score (DAS)28 at each evaluation visit. | 24 Weeks
The number of participants experiencing adverse events (AEs) as a measure of safety | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Scios, Inc. Clinical Trial, Study Director — Scios, Inc.